CLINICAL TRIAL: NCT00565747
Title: The Effect of Granulocyte-macrophage Colony Stimulating Factor (GM-CSF) During in Vitro Culture of Human Embryos on Subsequent Implantation Rates.
Brief Title: Efficacy Study of Granulocyte-macrophage Colony Stimulating Factor (GM-CSF) for Use in Human IVF
Acronym: GM-CSF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Origio A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DK001; Journal no. 8313-24 (Other: Danish Medicines Agency); Journal no. 461:2007/78029 (Other: Medical Products Agency - Sweden)
Record Dates: First submitted 2007-11-28; First posted 2007-11-30 (Estimated); Results first posted 2013-11-08 (Estimated); Last update posted 2015-05-15 (Estimated); Status verified 2015-04

CONDITIONS: Infertility
Keywords: GM-CSF; infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test culture (Experimental): Culture with GM-CSF
  Interventions: Device: Test culture
- Control culture (Placebo Comparator): Culture without GM-CSF
  Interventions: Device: Control culture

INTERVENTIONS:
Device: Test culture — A standard culture medium with added GM-CSF (ready-to-use)
  Other Names: EmbryoGen
  Arms: Test culture
Device: Control culture — The same standard culture medium, but without any additions (ready-to-use)
  Other Names: EmbryoAssist
  Arms: Control culture

SUMMARY:
This study is to assess whether addition of 2 ng/ml GM-CSF into a specific culture medium will increase the chance of a pregnancy after in vitro fertilisation.

DETAILED DESCRIPTION:
Throughout its development, the embryo is naturally exposed to a large number of cytokines and growth factors that are present in the woman's reproductive organs. A growing body of evidence indicates that these factors play a physiological role in the regulation of normal development of the pre-implanted embryo and that these factors therefore help to increase the implantation of the embryo and subsequently ensure optimal development of both foetus and placenta. The cytokine granulocyte-macrophage colony-stimulating factor (GM-CSF) has been shown to be present in the female reproductive organs during early pregnancy in mice, sheep, cows and humans.

2 ng/ml GM-CSF has been proven safe in a previous study presented at the European Society of Human Reproduction and Embrylogy (ESHRE) congress 2007 (A. Loft et al. 2007).

The present investigation (DK001) is to our knowledge the first large prospective randomised in vivo study in humans. Previous publications counting one Korean pilotstudy of 154 women prospectively randomised between culture medium with and without GM-CSF 2 ng/ml (Kim et al., 2001), showing a significant effect of GM-CSF on embryo implantation rate.

Based on this knowledge we hypothesize that culture of human embryos in the presence of GM-CSF will significantly increase the implantation rate also in a larger population.

This hypothesis is being tested by conducting a multicentre, randomised, parallel group, double-blind, placebo-controlled study with adaptive design, performed at 14 study centres. Each patient will participate in the study from retrieval of oocytes following standard hormonal treatment and until the 12th gestational week. Further a follow-up will be performed on pregnancies and children born.

The test group will include a standard culture medium with 2 ng/ml GM-CSF added from the time of insemination, and the control group will be the exact same medium but without any additions.

All procedures are according to standards of the clinic, with applied standard media except for the patient randomised study medium which is used for oocyte insemination, embryo culture and transfer. Embryo transfer will be performed Day 3.

An interim analysis has been performed for final sample size calculation.

ELIGIBILITY:
Inclusion Criteria:

* The couple or single woman has signed an informed consent form before any trial-related activities.
* In Vitro Fertilization (IVF) or IntraCytoplasmic Sperm Injection (ICSI) treatment indicated
* 25-39 years of age (both inclusive)
* Regular menstrual cycle: 21-35 days (both inclusive)
* Women treated with a standard Gonadotropin-Releasing Hormone (GnRH) agonist or antagonist protocol and a Follicle Stimulating Hormone (FSH) / human Menopausal Gonadotropin (hMG) starting dose between 100 and 300 IU daily.
* human Chorionic Gonadotropin (hCG) administration when the leading follicle has a calculated diameter of minimum 17 mm, or the day after.
* At least 3 follicles with a calculated diameter of ≥ 14 mm at the day of hCG.

Exclusion Criteria:

* The woman has previously participated in the DK001 study.
* Use of assisted hatching.
* Indication for Testicular Sperm Aspiration (TESA) or Percutaneous Epididymal Sperm Aspiration (PESA)
* Any medical conditions or genetic disorders prohibiting IVF/ICSI or interfering with the interpretation of results of the study (including pre-implantation genetic diagnostics).
* Use of any investigational drug within 30 days before oocyte retrieval
* Any severe chronic disease of relevance for reproductive function.
* Oocyte donation patients (donor or recipient).

Ages: 25 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1332 (Actual)
Dates: Start 2007-11; Primary Completion 2010-11 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Søren Ziebe, M.Sc., Principal Investigator — Rigshospitalet, Fertilitetsklinikken afd. 4071
Locations (14):
- Denmark (11):
  - Maigaard Fertilitetsklinik, Aarhus
  - Ciconia Aarhus Privathospital, Fertilitetsklinikken, Aarhus
  - Brædstrup Sygehus; IVF-Klinikken, Brædstrup
  - Rigshospitalet, Fertilitetsklinikken afd. 4071, Copenhagen
  - Fertilitetsklinikken Dronninglund, Dronninglund
  - IVF-SYD, Fredericia
  - Herlev Hospital, Fertilitetsklinikken G114F, Herlev
  - Holbæk Sygehus, Fertilitetsklinikken, Holbæk
  - Hvidovre Hospital; Fertilitetsklinikken afd. 455, Hvidovre
  - Odense Universitets Hospital, Fertilitetsklinikken, Odense
  - Regionshospitalet Skive, Fertilitetsklinikken, Skive
- Sweden (3):
  - IVF Kliniken Öresund, Malmo
  - Karolinska Universitetssjukhuset Huddinge, Fertilitetsenheten K59, Stockholm
  - Reproduktionscentrum, Uppsala

REFERENCES:
- [Derived] Rodriguez-Wallberg KA, Munding B, Ziebe S, Robertson SA. GM-CSF does not rescue poor-quality embryos: secondary analysis of a randomized controlled trial. Arch Gynecol Obstet. 2020 May;301(5):1341-1346. doi: 10.1007/s00404-020-05532-3. Epub 2020 Apr 9. PMID 32274634
- [Derived] Ziebe S, Loft A, Povlsen BB, Erb K, Agerholm I, Aasted M, Gabrielsen A, Hnida C, Zobel DP, Munding B, Bendz SH, Robertson SA. A randomized clinical trial to evaluate the effect of granulocyte-macrophage colony-stimulating factor (GM-CSF) in embryo culture medium for in vitro fertilization. Fertil Steril. 2013 May;99(6):1600-9. doi: 10.1016/j.fertnstert.2012.12.043. Epub 2013 Feb 4. PMID 23380186

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall recruitment period: October 2007 until August 2010. Patients were recruited at both public and private IVF clinics
Pre-assignment Details: Patients with informed consent but where it turned out that the inclusion/exclusion criteria were not fulfilled before assignment to groups, were excluded from the per-protocol (PP) analysis.
Groups:
- Test Culture: Culture with 2 ng/ml GM-CSF
Period: Overall Study
Arm/Group | Test Culture | Control Culture
Started | 654 | 678
Completed | 587 (Completed with an embryo transfer) | 605 (Completed with an embryo transfer)
Not Completed | 67 | 73
Not completed — No embryo transfer | 67 | 73

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test Culture | Control Culture | Total
Number analyzed (Participants) | 654 | 678 | 1332
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.2 (3.7) | 32.4 (3.8) | 32.3 (3.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 654 | 678 | 1332
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Denmark | 610 | 635 | 1245
  Sweden | 44 | 43 | 87

OUTCOME MEASURES:

1. Primary Outcome: Ongoing Implantation Rate Week 7
Description: Defined as number of gestational sacs with fetal heart beat, shown by ultrasound in gestational week 7 in percentage of number of embryo transferred.
Time Frame: Approximately 5 weeks from oocyte pick-up (corresponding to 7 weeks from ovulation)
Population: PP-population
Measure: Number; unit: percentage of transferred embryos
Units Other Than Participants: Embryos transferred
Arm/Group | Test Culture | Control Culture
Number analyzed (Participants) | 564 | 585
Number analyzed (Embryos transferred) | 838 | 882
percentage of transferred embryos | 23.5 | 20.0

2. Secondary Outcome: Number of Top Quality Embryos (TQE´s)
Description: Number of 4-5 cell embryo at 44 hours,at least 7 cell embryo at 68 hours, maximum 20% fragmentation, equally large blastomeres (less than 25% difference in size),No signs of multinucleation. Calculated in percentage of number of 2 pronuclei (2PN) oocytes.
Time Frame: 3 days from oocyte pick-up
Population: PP-population
Measure: Number; unit: percentage of 2PN's
Arm/Group | Test Culture | Control Culture
Number analyzed (Participants) | 564 | 585
percentage of 2PN's | 15.6 | 16.8

3. Secondary Outcome: Live Birth
Description: Subject having at least one live birth. Including a foetus which breathes or shows any other evidence of life after expulsion/extraction from its mother. The definition is independent of the duration of the pregnancy (ICMART/WHO criteria).
Time Frame: Until 7 days after birth
Population: PP-population
Measure: Number; unit: percentage of transfer patients
Arm/Group | Test Culture | Control Culture
Number analyzed (Participants) | 564 | 585
percentage of transfer patients | 28.9 | 24.1

ADVERSE EVENTS:
Arm/Group | Test Culture | Control Culture
Serious Adverse Events (participants affected / at risk) | 13/654 | 8/678
Other Adverse Events (participants affected / at risk) | 6/654 | 6/678
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Culture (N=654) | Control Culture (N=678)
Abdominal haemorrhage after oocyte pick-up. (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Ovarian Hyperstimulation Syndrome (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Uterine retension, haematuria and cystitis (General disorders) | 0 (0) | 1 (1)
Ovarian torsion (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Ectopic pregnancy (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Miscarriage (missed abortion) (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 1 (1)
Foetus or child born with malformations (General disorders) | 4 (4) | 4 (4)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Culture (N=654) | Control Culture (N=678)
Miscarriage (Pregnancy, puerperium and perinatal conditions) | 6 (6) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Confidentiality until publication of the main results of the study